CLINICAL TRIAL: NCT03056209
Title: A Dose Block-randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation, Phase I Clinical Study
Brief Title: Safety, Tolerability and Pharmacokinetic Study of KL1333 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KL1333_101
Record Dates: First submitted 2017-02-05; First posted 2017-02-17 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: MELAS Syndrome; Mitochondrial Respiratory Chain Deficiencies
Keywords: Mitochondrial DNA tRNALeu(UUR) m.3243A<G Mutation
MeSH Terms: conditions — MELAS Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- KL1333 25mg (Experimental): Group 1
  Interventions: Drug: KL1333 25 mg; Drug: Placebo
- KL1333 50mg (Experimental): Group 2
  Interventions: Drug: KL1333 50 mg; Drug: Placebo
- KL1333 100mg (Experimental): Group 3
  Interventions: Drug: KL1333 100 mg; Drug: Placebo
- KL1333 200mg (Experimental): Group 4
  Interventions: Drug: KL1333 200 mg; Drug: Placebo
- KL1333 400mg (Experimental): Group 5
  Interventions: Drug: KL1333 400 mg; Drug: Placebo
- KL1333 600mg (Experimental): Group 6
  Interventions: Drug: KL1333 600 mg; Drug: Placebo
- KL1333 800mg (Experimental): Group 7
  Interventions: Drug: KL1333 800 mg; Drug: Placebo

INTERVENTIONS:
Drug: KL1333 25 mg — oral administration, single dose, 25 mg 1 tab
  Arms: KL1333 25mg
Drug: KL1333 50 mg — oral administration, single dose, 25 mg 2 tabs
  Arms: KL1333 50mg
Drug: KL1333 100 mg — oral administration, single dose, 100 mg 1 tab
  Arms: KL1333 100mg
Drug: KL1333 200 mg — oral administration, single dose, 100 mg 2 tabs
  Arms: KL1333 200mg
Drug: KL1333 400 mg — oral administration, single dose, 100 mg 4 tabs
  Arms: KL1333 400mg
Drug: KL1333 600 mg — oral administration, single dose, 100 mg 6 tabs
  Arms: KL1333 600mg
Drug: KL1333 800 mg — oral administration, single dose, 100 mg 8 tabs
  Arms: KL1333 800mg
Drug: Placebo — oral administration, placebo

SUMMARY:
The purpose of this First In Human study is to investigate the safety and tolerability of KL1333 after a single oral dose and to investigate the pharmacokinetic characteristics of KL1333 after a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* 19 - 45 years of age at the time of screening
* Subjects weighing ≥55 and ≤90 kg with BMI between 18 and 27 kg/m2
* Subjects who agreed to voluntarily participate in this study and comply with all the study requirements by signing informed consent form after being informed of the nature of this study and understanding all aspects of this study

Exclusion Criteria:

* History of clinically significant hepatic, renal, neurologic, immunologic, respiratory, endocrine disease or hematologic•oncologic disease, cardiovascular, psychiatric disease
* History of disease or surgery of the gastrointestinal tract that could interfere with kinetics of the study drug. Simple hernia repair or appendectomy are excepted.
* History of clinically significant or relevant allergy/hypersensitivity
* Blood AST (SGOT), ALT (SGPT) >1.5 of upper limit
* eGFR value of ≤90mL/min/1.73m2
* Systolic blood pressure of <100 mmHg or >160 mmHg
* Diastolic blood pressure of <60 mmHg or >100 mmHg
* Any abnormalities in 12-lead ECG at screening visit
* Subjects who showed positive result in drug abuse tests, or who has history of drug abuse within 60 days prior to the time of screening
* Subjects who took prescribed medications or oriental medicine within 14 days or over-the-counter (OTC) medications or vitamins within 7 days prior to the dose of the study drug (however, the subject can be included if other criteria are met according to the discretion of the investigator)
* Subjects who were administered any investigational products within 3 months from the first dose of the study drug
* Subjects who have donated whole blood (60 days) or partial blood (30 days), or received blood transfusion
* Subjects who have had alcohol consistently (>21units/week, 1unit=10 g of pure alcohol) or who is not able to stop drinking alcohol throughout the study period
* Subjects who have smoked until 90 days prior to the study initiation or who are not able to stop smoking throughout the study period
* Subjects who are not able to stop taking grapefruit/caffeine from 3 days prior to the first dose of the study drug throughout the study period
* Subjects who plan for pregnancy during the study period or who are not able to use established contraceptive method
* Subject who judged not eligible for study participation by investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Number of reported adverse events | from day 1 to day 15

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of KL1333 | from day 1 to day 15
Area Under the Curve (AUC) of KL1333 | from day 1 to day 15
Half-life (T1/2) of KL1333 | from day 1 to day 15

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD., MBA, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No